CLINICAL TRIAL: NCT04881864
Title: Adapting an Evidence-Based Exercise Program for Remote Delivery to Rural Older Adults
Brief Title: Study for Rural Innovations in the Delivery of Exercise
Acronym: STRIDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kushang Patel, Research Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00011517
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis
Keywords: Physical Activity; Rural; Older Adults
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-EF (Experimental): Livestream, instructor-led tele-exercise classes, involving balance, endurance, and strength training
  Interventions: Behavioral: Tele-Enhance Fitness

INTERVENTIONS:
Behavioral: Tele-Enhance Fitness — Livestream, instructor-led tele-exercise classes, involving balance, endurance, and strength training

SUMMARY:
: Falls are the primary cause of injury and a leading cause of disability and mortality among older adults. Risk factors for falling are common among older adults with knee osteoarthritis (OA) - a highly prevalent condition. Physical exercise is consistently the most efficacious intervention for preventing falls in older adults. However, access to these programs is severely limited in rural settings. Considering that rural communities have a higher disease burden and higher proportion of older adults than non-rural areas, there is a critical need to (1) adapt evidence-based exercise programs for remote delivery to increase access for rural older adults and (2) develop pathways to implement exercise programs in rural health care systems that consistently reach and engage patients with knee OA. Accordingly, the proposed project aims to refine a protocol for remote delivery of Enhance Fitness (EF). EF is an evidence-based, group exercise program involving strength, endurance, and balance training that is recommended for falls prevention and OA management

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* English-speaking
* Physician diagnosed knee osteoarthritis
* Knee pain that occurs almost daily for at least the past 3 months and is moderate to severe in intensity
* Knee pain-related difficulty with walking or climbing stairs
* resident of a rural county

Exclusion Criteria:

* cognitive impairment determined by a Mini Montreal Cognitive Assessment score of <11
* any of the following in the past 6 months: cancer requiring treatment (except for non- melanoma skin cancer), heart attack, stroke, hip fracture, hip/knee replacement, spinal surgery, heart surgery, deep vein thrombosis, or pulmonary embolus; and temporary exclusions
* hospitalization within the last month
* ≥3 falls within the past month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability of Tele-Enhance Fitness | 12 weeks
  Feasibility outcomes include intervention engagement and adherence, retention, fidelity of tele-EF treatment, and adverse events. Multiple dimensions of acceptability will be assessed from qualitative interviews with participants and instructors.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function 8-item Short Form | Change from baseline PROMIS physical function score at 12 weeks
  Patient-reported physical functioning
Knee injury and Osteoarthritis Outcome Score (KOOS) Physical Function Subscale | Change from Baseline KOOS Physical Function Subscale score at 12 weeks
  Patient-reported knee pain-related interference with physical functioning

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators recognize that data sharing leads to the promotion of science. We intend to publish the results of the proposed study and will make data available to investigators upon request (following publication). The final dataset will include demographic, clinical, and behavioral data on 15 older adults followed over a 3-month period. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that the possibility of deductive disclosure of subjects with unusual characteristics remains. For these reasons, we propose to make the data and associated documentation available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.